CLINICAL TRIAL: NCT03249701
Title: Electrical Acupoint Stimulation for Postoperative Recovery After Knee Arthroplasty. A Randomized, Double-blind, Clinical Trial.
Brief Title: Electrical Acupoint Stimulation for Postoperative Recovery
Acronym: EAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, weiliang zhang, Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SZH-A-20170501-R2
Record Dates: First submitted 2017-08-03; First posted 2017-08-15 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Postoperative Complications; Postoperative Nausea and Vomiting; Postoperative Infection; Postoperative Delirium; Postoperative Pneumonia; Deep Vein Thrombosis; Postoperative Retention of Urine; Postoperative Recovery
Keywords: Acupoint Stimulation; postoperative recovery; Postoperative Complications; Peri-operation
MeSH Terms: conditions — Postoperative Complications; Postoperative Nausea and Vomiting; Emergence Delirium; Venous Thrombosis | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: The participants divided into 3 groups randomized, one group receive transcutaneous electrical acupoint stimulation, one group receive electroacupuncture, the third group only connect to acupoints without stimulation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The intervention administered randomly to the participants. The participants, care providers, investigator, outcomes assessor done their job, separately. The blind will be controlled by a assigned investigator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEAS group (Experimental): Transcutaneous Electrical Acupoint Stimulation on Neiguan, Quchi, Zusanli, Sanyinjiao. Intensity: maximal tolerance by subject; Time span: 30minutes before anesthesia induction and 30 minutes after wound closure.
  Interventions: Device: Transcutaneous Electrical Acupoint Stimulation
- Electroacupuncture group (Placebo Comparator): Hand-needle on Neiguan, Quchi, Zusanli, Sanyinjiao.Intensity: maximal tolerance by subject; Time span: 30minutes before anesthesia induction and 30 minutes after wound closure.
  Interventions: Device: Electroacupuncture
- sham TEAS group (Sham Comparator): Sham transcutaneous electrical acupoint stimulation on Neiguan, Quchi, Zusanli, Sanyinjiao; Intensity: maximal tolerance by subject; Time span: 30minutes before anesthesia induction and 30 minutes after wound closure.
  Interventions: Device: sham Transcutaneous Electrical Acupoint Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Acupoint Stimulation — The intervention will be administered by electrical acupoint machine, the brand is Great Wall.
  Arms: TEAS group
Device: Electroacupuncture — The intervention will be administered by electrical acupoint machine, the brand is Great Wall.
  Arms: Electroacupuncture group
Device: sham Transcutaneous Electrical Acupoint Stimulation — The intervention will be administered by transcutaneous electrical acupoint machine, even no truly actualized.
  Arms: sham TEAS group

SUMMARY:
This study investigates electrical acupoint stimulation (EAS) administered in peri-operation for improving postoperative recovery in elder patients, who accept knee arthroplasty. the surgery cause to change of stress response, which might be associated with postoperative recovery of patient Totally, three groups are created, 1/3 participants receive transcutaneous electrical acupoint stimulation, 1/3 participants receive electroacupuncture, the rest 1/3 will use sham transcutaneous electrical acupoint stimulation.

DETAILED DESCRIPTION:
Theoretically, the application of electrical acupoint stimulation (EAS) base on the theory of traditional Chinese medicine. It deems that a surgery might consume Qi, then cause to imbalance of Qi and Blood, especially in elder patients. Besides, surgery lead to change of stress response (hormones). The EAS administration intra-operatively perhaps be beneficial to recovery of patients, reduce the incidence of postoperative complications. The main possible mechanism was stress response regulation. The hypothesis is that the EAS improve postoperative recovery of patient through regulating stress response.

ELIGIBILITY:
Inclusion Criteria:

* Agree to sign the contract
* The patients receive total hip or knee arthroplasty
* Epidural anesthesia administered

Exclusion Criteria:

* The patients' age out of range setting
* Forbidden to the administration of transcutaneous electrical acupoint stimulation
* Communication disorder
* The patients who had medical history of cerebral vascular diseases, deep vein thrombosis, urinary retention, nausea and vomiting.
* The patients who attended another trial in the past three months
* Emergency surgery

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
The postoperative recovery | 7 days
  Record the postoperative recovery after surgery through quality of recovery-40 questionnaire.

SECONDARY OUTCOMES:
The adverse event | 7 days
  Record all the adverse events appeared during the entire trail, which might cause to skin rash, allergic reaction, et al.
The level of stress response | up to 7 days
  Assess the level of preoperative stress response at 1, 3, 7 days after operation. It mainly include Adrenocorticotropic Hormone (ACTH), Cortisol (COR), Adrenaline (E), norepinephrine (NE). All measures unit is pg/ml.
Postoperative complications | 7 days
  Record the incidence of any postoperative complications during 7 days
The level of inflammatory response by TNF-a, IL-1, IL-6, IL-10 | up to 7 days
  Assess the level of perioperative inflammatory response at 1, 3, 7 days after operation. It mainly include Tumor Necrosis Factor-a (TNF-a), Interleukins-1 (IL-1), Interleukins-6 (IL-6), Interleukins-10 (IL-10). All measures unit is ng/ml.
The level of inflammatory response by C-reactive protein | up to 7 days
  Assess the level of perioperative inflammatory response at 1, 3, 7 days after operation through C-reactive protein. the unit is mg/L.

OTHER OUTCOMES:
Age in years | 1 day
  Once patients enrolled, the age (years) need to be recorded ahead of operation.
ASA classification status | 1 day
  Once patients enrolled, the ASA condition need to be recorded ahead of operation depend on the ASA classification.
Gender | 1 day
  Once patients enrolled, the gender need to be recorded ahead of operation.
Weight in kilograms | 1 day
  Once patients enrolled, the weight (kilograms) need to be recorded ahead of operation.
Height in meters | 1 day
  Once patients enrolled, the height (meters) need to be recorded ahead of operation.
BMI in kg/m^2 | 1 day
  Once patients enrolled, the BMI (weight and height will be combined to report BMI in kg/m^2) will be reported base on weight and height ahead of operation.

CONTACTS AND LOCATIONS:
Overall Officials: Su Fan, MD, Principal Investigator — Affiliated Hospital of Shandong University of Traditional Chinese Medicine
Locations (1):
- Affiliated hospital of shandong university of traditional chinese medicine, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
IPD sharing content included the intervention protocol, record or data collected for the primary and secondary outcome measures.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion, forever.
Access Criteria: Anyone are available to access the data collected on this website with requiring to sign the Data Access Agreement.

REFERENCES:
- [Result] Coburn M, Fahlenkamp A, Zoremba N, Schaelte G. Postoperative cognitive dysfunction: Incidence and prophylaxis. Anaesthesist. 2010 Feb;59(2):177-84; quiz 185. doi: 10.1007/s00101-009-1657-2. PMID 20084351
- [Result] Choi JB, Shim YH, Lee YW, Lee JS, Choi JR, Chang CH. Incidence and risk factors of postoperative nausea and vomiting in patients with fentanyl-based intravenous patient-controlled analgesia and single antiemetic prophylaxis. Yonsei Med J. 2014 Sep;55(5):1430-5. doi: 10.3349/ymj.2014.55.5.1430. PMID 25048507
- [Result] Office of the Surgeon General (US); National Heart, Lung, and Blood Institute (US). The Surgeon General's Call to Action to Prevent Deep Vein Thrombosis and Pulmonary Embolism. Rockville (MD): Office of the Surgeon General (US); 2008. Available from http://www.ncbi.nlm.nih.gov/books/NBK44178/ PMID 20669525
- [Result] Montazeri AS, Hamidzadeh A, Raei M, Mohammadiun M, Montazeri AS, Mirshahi R, Rohani H. Evaluation of Oral Ginger Efficacy against Postoperative Nausea and Vomiting: A Randomized, Double - Blinded Clinical Trial. Iran Red Crescent Med J. 2013 Dec;15(12):e12268. doi: 10.5812/ircmj.12268. Epub 2013 Dec 5. PMID 24693389
- [Result] Sorrell JM. Postoperative cognitive dysfunction in older adults: a call for nursing involvement. J Psychosoc Nurs Ment Health Serv. 2014 Nov;52(11):17-20. doi: 10.3928/02793695-20141021-03. PMID 25375388
- [Result] Ge Y, Ma Z, Shi H, Zhao Y, Gu X, Wei H. [Incidence and risk factors of postoperative cognitive dysfunction in patients underwent coronary artery bypass grafting surgery]. Zhong Nan Da Xue Xue Bao Yi Xue Ban. 2014 Oct;39(10):1049-55. doi: 10.11817/j.issn.1672-7347.2014.10.011. Chinese. PMID 25355258
- [Result] Tsay SL, Cho YC, Chen ML. Acupressure and Transcutaneous Electrical Acupoint Stimulation in improving fatigue, sleep quality and depression in hemodialysis patients. Am J Chin Med. 2004;32(3):407-16. doi: 10.1142/S0192415X04002065. PMID 15344424
- [Result] Kabalak AA, Akcay M, Akcay F, Gogus N. Transcutaneous electrical acupoint stimulation versus ondansetron in the prevention of postoperative vomiting following pediatric tonsillectomy. J Altern Complement Med. 2005 Jun;11(3):407-13. doi: 10.1089/acm.2005.11.407. PMID 15992223
- [Result] Yao Y, Zhao Q, Gong C, Wu Y, Chen Y, Qiu L, Wu X, Chen Y. Transcutaneous Electrical Acupoint Stimulation Improves the Postoperative Quality of Recovery and Analgesia after Gynecological Laparoscopic Surgery: A Randomized Controlled Trial. Evid Based Complement Alternat Med. 2015;2015:324360. doi: 10.1155/2015/324360. Epub 2015 Jun 11. PMID 26170873
- [Result] Zheng LH, Sun H, Wang GN, Liang J, Wu HX. Effect of transcutaneous electrical acupoint stimulation on nausea and vomiting induced by patient controlled intravenous analgesia with tramadol. Chin J Integr Med. 2008 Mar;14(1):61-4. doi: 10.1007/s11655-007-9006-2. PMID 18219451

DOCUMENTS (2):
  • Informed Consent Form (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03249701/ICF_002.pdf
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT03249701/Prot_SAP_003.pdf